CLINICAL TRIAL: NCT05142657
Title: Are There Dietary Factors Affecting the Development of Pancreatitis in Patients With Gallstones?
Status: Completed | Type: Observational
Sponsor: Istanbul Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Ufuk Oguz Idiz, Assoc. Prof. MD. PhD, Istanbul Training and Research Hospital
Other Study IDs: Pancreatitis diet
Record Dates: First submitted 2021-11-21; First posted 2021-12-02 (Actual); Last update posted 2022-04-14 (Actual); Status verified 2021-11

CONDITIONS: Diet Habit; Gall Stone; Pancreatitis
Keywords: meat; egg; fat; protein
MeSH Terms: conditions — Feeding Behavior; Gallstones; Pancreatitis; Platelet Glycoprotein IV Deficiency | interventions — Diet Surveys

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 7 Days
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Case: Patients who have gallstone pancreatitis
  Interventions: Other: diet survey
- Control: Patients who have only gallstone
  Interventions: Other: diet survey

INTERVENTIONS:
Other: diet survey — Dietary survey applied to all participants

SUMMARY:
The most common cause of acute pancreatitis is gallstones. It is known that diet and obesity play a role in the formation of gallstones. It has been reported that the risk of gallstone formation is two times higher in obese individuals with a body mass index (BMI) >30 than in normal-weight individuals with a BMI between 20-25. The epidemiological literature on the relationship between diet and risk of acute pancreatitis is very limited. In addition, it is often unclear which type (acute, recurrent, or chronic) and subtype (gallstone-related or non-gallstone-related) of acute pancreatitis is studied in studies. Although there are studies in the literature evaluating the relationship between diet and development of gallstones or the development of pancreatitis with diet, studies examining the role of diet in the development of pancreatitis in patients with gallstones are very limited. In this study, we aimed to investigate the dietary differences in patients with gallstones who had pancreatitis and those who did not.

DETAILED DESCRIPTION:
The incidence of acute pancreatitis has been reported as 4.9-35/100.000, and the incidence increases every year with the increase in obesity and gallstone rates. It is most commonly observed between the ages of 30-60 and no difference was found in terms of gender distribution. The most common cause of acute pancreatitis is gallstones. Alcohol use, drugs and other reasons come next.

It is known that diet and obesity play a role in the formation of gallstones. It has been reported that the risk of gallstone formation is two times higher in obese individuals with a body mass index (BMI) >30 than in normal-weight individuals with a BMI between 20-25. In addition, many studies have reported that increased use of dietary refined carbohydrates and triglycerides and reduced dietary fiber intake are associated with gallstone formation.

The epidemiological literature on the relationship between diet and risk of acute pancreatitis is very limited. In addition, it is often unclear which type (acute, recurrent, or chronic) and subtype (gallstone-related or non-gallstone-related) of acute pancreatitis is studied in studies. On the other hand, Sarles et al. In a comprehensive study conducted in 1973, he reported that high fat and protein consumption and alcoholism increase the risk of pancreatitis, regardless of etiology. Few case-control and ecological studies have evaluated the effect of protein, fat, and carbohydrate intakes on alcohol-related or gallstone-related acute pancreatitis risk or non-gallstone-related acute pancreatitis risk or acute pancreatitis mortality.

At the beginning of the twentieth century, an inverse relationship between coffee consumption and the risk of alcohol-induced acute pancreatitis was observed in a prospective study, and an inverse relationship with fruit consumption in two smaller case-control studies, and a positive association with consumption of freshwater fish and parboiled rice. In parallel, overly large meals and food allergies after a long period of fasting have been reported to be risk factors for acute pancreatitis.

Although there are studies in the literature evaluating the relationship between diet and development of gallstones or the development of pancreatitis with diet, studies examining the role of diet in the development of pancreatitis in patients with gallstones are very limited. In this study, we aimed to investigate the dietary differences in patients with gallstones who had pancreatitis and those who did not.

In the study, age, gender, body mass index, alcohol and cigarette consumption status, daily physical activity status, eating frequency, frequency of food consumption for three days, and their food consumption status will be evaluated with the BeBis 8 Full version program and it will be compared whether there is a difference between patients who had pancreatitis and those who did not. .

ELIGIBILITY:
Inclusion criteria in the pancreatitis group were :

* 18-80 years of age,
* having gallbladder stones
* being diagnosed with pancreatitis, exclusion criteria in the pancreatitis group were:
* having any cancer,
* being pregnant,
* having chronic liver or kidney disease,
* icterus,
* developing after ERCP.

Inclusion criteria in the control group were:

* 18-80 years of age
* gallbladder stones, exclusion criteria in the control group were:
* any cancer,
* pregnancy,
* chronic liver or kidney disease,
* icterus,
* previous pancreatitis attack

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All the participants have gallstone. In control group participants did not have any pancreatitis history. In case group patients have pancreatitis.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2021-11-20 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
energy, cholesterol, protein, fat | 3 days
  Daily energy, cholesterol, protein, fat intake of the participants

CONTACTS AND LOCATIONS:
Overall Officials: Ufuk O İdiz, M.D, Principal Investigator — Istanbul Training and Research Hospital
Locations (1):
- Istanbul Traininng and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Setiawan VW, Pandol SJ, Porcel J, Wei PC, Wilkens LR, Le Marchand L, Pike MC, Monroe KR. Dietary Factors Reduce Risk of Acute Pancreatitis in a Large Multiethnic Cohort. Clin Gastroenterol Hepatol. 2017 Feb;15(2):257-265.e3. doi: 10.1016/j.cgh.2016.08.038. Epub 2016 Sep 5. PMID 27609706
- [Background] Dugum M, Gougol A, Paragomi P, Gao X, Matta B, Yazici C, Tang G, Greer P, Pothoulakis I, O'Keefe SJD, Whitcomb DC, Yadav D, Papachristou GI. Association of Dietary Habits with Severity of Acute Pancreatitis. Curr Dev Nutr. 2018 Oct 8;2(12):nzy075. doi: 10.1093/cdn/nzy075. eCollection 2018 Dec. PMID 30569031